CLINICAL TRIAL: NCT05415696
Title: Prostatic Artery Embolization (PAE) for the Treatment of Lower Urinary Tract Symptoms (LUTS) in Prostate Cancer Patients Undergoing Radiation Therapy
Brief Title: Prostatic Artery Embolization for the Treatment of Lower Urinary Tract Symptoms in Prostate Cancer Patients Undergoing Radiation Therapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrolling to this clinical trial was too difficult
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Andrew Picel, Clinical Associate Professor, Radiology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-64391; PROS0108 (Other: Stanford OnCore)
Record Dates: First submitted 2022-06-08; First posted 2022-06-13 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Prostate Cancer
Keywords: Prostatic artery embolization; Lower urinary tract symptoms
MeSH Terms: conditions — Prostatic Neoplasms; Lower Urinary Tract Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prostatic artery embolization (PAE) (Other): Study participants will be treated with a single PAE procedure performed with Embosphere microspheres.
  Interventions: Procedure: Prostatic artery embolization

INTERVENTIONS:
Procedure: Prostatic artery embolization — Patients will undergo PAE with 100-300 µm or 300-500 µm Embospheres following standard PAE technique performed by Interventional Radiology at Stanford University

SUMMARY:
The purpose of this study is to learn if the prostatic artery embolization procedure can reduce urinary tract symptoms in patients with enlarged prostates and prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE

1. To evaluate the symptomatic improvement in lower urinary tract symptoms after prostatic artery embolization (PAE)

SECONDARY OBJECTIVES

1. To evaluate objective measures of improved urinary obstruction after PAE: urine flow rate, prostate volume, and post-void residual
2. To measure effects of PAE on prostate specific antigen (PSA).
3. To evaluate if PAE reduces the prostate volume and simplifies radiation therapy
4. To evaluate the safety of PAE performed in this patient population

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years and ≤ 90 years old
* Prostate volume ≥ 40 mL and ≤ 300 mL
* Biopsy proven prostate cancer undergoing radiation therapy
* Diagnosis of moderate to severe lower urinary tract symptoms (LUTS) defined as at least one of the following:

  1. IPSS ≥ 12 or dependent on urinary catheterization, or
  2. IPSS Quality of Life (QoL) assessment ≥ 3, and
  3. Qmax ≤ 12 mL/sec
* Ability to understand and willingness to sign the written consent

Exclusion Criteria:

* Neurogenic bladder disorder due to multiple sclerosis, Parkinson's disease, spinal cord injury, diabetes, etc., as demonstrated on urodynamic testing.
* Detrusor muscle failure, urethral stenosis, or urinary obstruction due to causes other than prostatic obstruction, as demonstrated on urodynamic testing
* Bladder diverticula greater than 5 cm or bladder stones greater than 2 cm
* Other active urogenital cancer
* Baseline serum creatinine greater than 2 mg/dL
* Evidence of tortuous or atherosclerotic blood vessels
* Coagulation disturbances not normalized by medical treatment
* Allergy to iodinated contrast agents not responsive to steroid premedication regimen

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09-19 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in symptom score using the International Prostate Symptom Scale (IPSS) | 2 months
  Patients will be classified into one of 3 symptom severity categories based on their total IPSS score as follows:
  Mildly symptomatic: 0-7 Moderately symptomatic: 8-19 Severely symptomatic: 20-35

SECONDARY OUTCOMES:
Mean change from baseline in maximal urinary flow measured | at baseline, 2 months, and 12 months after intervention
Mean change from baseline in post-void residual measured | at baseline, 2 months, and 12 months after intervention
Mean change from baseline in prostate volume measure | at baseline, 2 months, and 12 months after intervention
Mean change from baseline in international prostate symptom scale to measure long term subjective outcomes measured | at baseline, 2 months, and 12 months after intervention
  Patients will be classified into one of 3 symptom severity categories based on their total IPSS score as follows:
  Mildly symptomatic: 0-7 Moderately symptomatic: 8-19 Severely symptomatic: 20-35
Mean change from baseline prostate specific antigen measure | at baseline, 2 months, and 12 months after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Picel, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Cancer Center, San Francisco, California, United States